CLINICAL TRIAL: NCT05948202
Title: Impact of Mindfulness-Enhanced Pivotal Response Group Treatment on Parenting Stress: A Randomized Controlled Trial
Brief Title: Mindfulness-Enhanced Pivotal Response Group Treatment on Parenting Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Angela Scarpa-Friedman, Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-079
Record Dates: First submitted 2023-06-01; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mPRT (Experimental): mindfulness-enhanced Pivotal Response Treatment: group pivotal response training for parents that is supplemented with mindfulness strategies
  Interventions: Behavioral: Pivotal Response Treatment
- pPRT (Active Comparator): psychoeducation-enhanced Pivotal Response Treatment: group pivotal response training for parents that is supplemented with psychoeducation about stress and stress reduction
  Interventions: Behavioral: Pivotal Response Treatment

INTERVENTIONS:
Behavioral: Pivotal Response Treatment — Group-based parent training to teach parents behavioral strategies based on principles of learning to motivate their child.

SUMMARY:
This project tests the feasibility and preliminary proof of concept for a mindfulness-enhanced adaptation of Pivotal Response Treatment on parenting stress and child communication, using a randomized controlled design.

DETAILED DESCRIPTION:
One of the core features of Autism Spectrum Disorder (ASD), social communication impairment, presents in a variety of ways, including reduced functional language use and social initiations, which often warrant intensive intervention services. Additionally, parents of children with ASD demonstrate increased levels of parenting stress when compared to parents of typically developing children and children with developmental delays. Elevated parenting stress has been shown to diminish positive treatment outcomes, which lends support to develop methodologies to concomitantly target child and parent behaviors. The current randomized control trial (RCT) uses a dual-pronged approach to directly target both child communication deficits and parenting stress within a group format. This RCT combined an empirically supported behavioral therapy, Pivotal Response Treatment (PRT), with components from Acceptance and Commitment Therapy and Mindful Parenting for reducing parenting stress. Caregivers and their minimally or pre-verbal child with diagnosed or suspected ASD were randomly assigned to one of the following supplemental conditions: mindfulness-enhanced PRT (mPRT) or psychoeducation-enhanced PRT (pPRT) as an active control condition. The current study assessed feasibility and acceptability in addition to demonstrating proof of concept in regard to additive effects of mPRT compared to pPRT.

ELIGIBILITY:
Inclusion Criteria:

* For children: minimally verbal or nonverbal, 1.5 to 6 years old, current or suspected autism spectrum disorder diagnosis, demonstrated ability to make meaningful vocalizations
* For parents: willingness to attend group treatment sessions, record weekly videos, and share videos in a group setting

Exclusion Criteria:

* For children, no active medical problems (e.g., unstable seizure disorders)
* For parents, no severe mental health problems (e.g., suicidal intent, psychosis)

Ages: 18 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2020-02-04 (Actual)

PRIMARY OUTCOMES:
Therapist fidelity observation | weekly, from start of treatment through 12 weeks
  observation at 30-second intervals; number out of 10 pivotal response therapy components observed for each 30-second interval of the recording and then averaged over the length of the recording (which were 5-10 minutes long)
Child utterances - observation | pre-treatment at intake
  level or amount of child utterances during a structured laboratory task observation
Child utterances - observation | mid-treatment, at 6 weeks from start of treatment
  level or amount of child utterances during a structured laboratory task observation
Child utterances - observation | weekly, from start of treatment through 12 weeks
  level or amount of child utterances during a structured laboratory task observation
Child utterances - observation | post-treatment, at 12 weeks from start of treatment
  level or amount of child utterances during a structured laboratory task observation
Child utterances - observation | follow-up, at 3 months after the last treatment session
  level or amount of child utterances during a structured laboratory task observation
Parent fidelity observation | weekly, from start of treatment through 12 weeks
  observation at 30-second intervals; number out of 10 pivotal response therapy components observed for each 30-second interval of the recording and then averaged over the length of the recording (which were 5-10 minutes long)
Parenting Stress Index, 4th edition | pre-treatment at intake
  level of parent-reported stress;
Parenting Stress Index, 4th edition | mid-treatment, at 6 weeks from start of treatment
  level of parent-reported stress
Parenting Stress Index, 4th edition | post-treatment, at 12 weeks from start of treatment
  level of parent-reported stress
Parenting Stress Index, 4th edition | follow-up, at 3 months after last treatment session
  level of parent-reported stress
Autism Parenting Stress Index | pre-treatment at intake
  level of parent-reported stress specific for parents of young autistic children
Autism Parenting Stress Index | mid-treatment, at 6 weeks from start of treatment
  level of parent-reported stress specific for parents of young autistic children
Autism Parenting Stress Index | post-treatment, at 12 weeks from start of treatment
  level of parent-reported stress specific for parents of young autistic children
Autism Parenting Stress Index | follow-up, at 3 months after last treatment session
  level of parent-reported stress specific for parents of young autistic children
Subjective Units of Parenting Stress Scale | pre-treatment at intake
  level of parent-reported stress immediately following the structured lab observation, with 0 signifying no stress and 100 signifying extreme stress
Subjective Units of Parenting Stress Scale | mid-treatment, at 6 weeks from start of treatment
  level of parent-reported stress immediately following the structured lab observation, with 0 signifying no stress and 100 signifying extreme stress
Subjective Units of Parenting Stress Scale | post-treatment, at 12 weeks from start of treatment
  level of parent-reported stress immediately following the structured lab observation, with 0 signifying no stress and 100 signifying extreme stress
Subjective Units of Parenting Stress Scale | follow-up, at 3 months after last treatment session
  level of parent-reported stress immediately following the structured lab observation

SECONDARY OUTCOMES:
Parent Feelings Questionnaire | pre-treatment, at intake
  parent-report of positive and negative feelings toward the child; 5 point scale from definitely untrue for me to definitely true for me; higher scores mean higher levels of the feeling
Parent Feelings Questionnaire | mid-treatment, at 6 weeks from start of treatment
  parent-report of positive and negative feelings toward the child; 5 point scale from definitely untrue for me to definitely true for me; higher scores mean higher levels of the feeling
Parent Feelings Questionnaire | post-treatment, at 12 weeks from start of treatment
  parent-report of positive and negative feelings toward the child; 5 point scale from definitely untrue for me to definitely true for me; higher scores mean higher levels of the feeling
Parent Feelings Questionnaire | follow-up, at 3 months after last treatment session
  parent-report of positive and negative feelings toward the child; 5 point scale from definitely untrue for me to definitely true for me; higher scores mean higher levels of the feeling
Positive and Negative Affect Schedule | pre-treatment, at intake
  parent-reported positive and negative affect in adults; 5 point scale from very slightly to extremely; higher scores mean higher levels of the feeling
Positive and Negative Affect Schedule | mid-treatment, at 6 weeks from start of treatment
  parent-reported positive and negative affect in adults; 5 point scale from very slightly to extremely; higher scores mean higher levels of the feeling
Positive and Negative Affect Schedule | post-treatment, at 12 weeks from start of treatment
  parent-reported positive and negative affect in adults; 5 point scale from very slightly to extremely; higher scores mean higher levels of the feeling
Positive and Negative Affect Schedule | follow-up, at 3 months after last treatment session
  parent-reported positive and negative affect in adults; 5 point scale from very slightly to extremely; higher scores mean higher levels of the feeling
Five Facet Mindfulness Questionnaire | pre-treatment, at intake
  parent-reported propensity toward mindfulness in everyday life; 5 point scale from never true to always true; higher scores mean more mindfulness
Five Facet Mindfulness Questionnaire | mid-treatment, at 6 weeks from start of treatment
  parent-reported propensity toward mindfulness in everyday life; 5 point scale from never true to always true; higher scores mean more mindfulness
Five Facet Mindfulness Questionnaire | post-treatment, at 12 weeks from start of treatment
  parent-reported propensity toward mindfulness in everyday life; 5 point scale from never true to always true; higher scores mean more mindfulness
Five Facet Mindfulness Questionnaire | follow-up, at 3 months after last treatment session
  parent-reported propensity toward mindfulness in everyday life; 5 point scale from never true to always true; higher scores mean more mindfulness
Acceptance and Action Questionnaire | pre-treatment, at intake
  parent-reported level of experiential avoidance, on a 7 point scale from never true to always true; higher scores indicate more avoidance
Child Behavior Checklist for ages 1.5 to 5 | mid-treatment, at 6 weeks from start of treatment
  parent-reported measure of child emotional and behavioral concerns; converted to t-scores; higher scores indicate higher levels of the behavior problem
Child Behavior Checklist for ages 1.5 to 5 | post-treatment, at 12 weeks from start of treatment
  parent-reported measure of child emotional and behavioral concerns; converted to t-scores; higher scores indicate higher levels of the behavior problem
Child Behavior Checklist for ages 1.5 to 5 | follow-up, at 3 months after last treatment session
  parent-reported measure of child emotional and behavioral concerns; converted to t-scores; higher scores indicate higher levels of the behavior problem

OTHER OUTCOMES:
Parent Treatment Satisfaction Questionnaire | post-treatment, at 12 weeks from start of treatment
  Parent-reported satisfaction with the treatment protocol on a 5 point scale from would not recommend to strongly recommend; not at all helpful to very helpful; not at all difficult to very difficult; and too few sessions to too many sessions.

CONTACTS AND LOCATIONS:
Locations (1):
- Virginia Tech Autism Clinic, Blacksburg, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data are shared with other members of the research team.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Hayes SA, Watson SL. The impact of parenting stress: a meta-analysis of studies comparing the experience of parenting stress in parents of children with and without autism spectrum disorder. J Autism Dev Disord. 2013 Mar;43(3):629-42. doi: 10.1007/s10803-012-1604-y. PMID 22790429
- [Background] Osborne LA, McHugh L, Saunders J, Reed P. Parenting stress reduces the effectiveness of early teaching interventions for autistic spectrum disorders. J Autism Dev Disord. 2008 Jul;38(6):1092-103. doi: 10.1007/s10803-007-0497-7. Epub 2007 Nov 20. PMID 18027079

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT05948202/Prot_SAP_000.pdf